CLINICAL TRIAL: NCT05508139
Title: The Role Of Vestibular Rehabilitation Therapy In Management Of Vestibular Migraine Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelmawla hammad abdelmawla kassem, The Role Of Vestibular Rehabilitation Therapy In Management Of Vestibular Migraine Patients, Assiut University
Other Study IDs: vestibular rehablitation
Record Dates: First submitted 2022-08-15; First posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Vestibular Migraine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. To assess the criteria of positional vertigo in vestibular migraine patients
2. To assess the effect of vestibular rehabilitation therapy in management of positional vertigo in vestibular migraine patients

DETAILED DESCRIPTION:
Vestibular migraine(VM) is a variant of migraine where the patient reports recurrent vertigo lasting minutes to days. The migraine headache component may be present with associated light and sound sensitivity but the vestibular symptoms are usually prominent . Migraine prophylaxis has been shown to provide some benefit to help to prevent or abort acute attacks of vertigo .

Vestibular migraine has a life time prevalence of about 1 % and a 1-year prevalence of 0.9 % in the general population and accounts for about 7% of patients seen in dizziness clinics and 9 % of patients seen in migraine clinics .

The International Headache Society and the International Barany Society for Neuro-otology have developed a consensus document with diagnostic criteria for VM . This diagnosis was included in the appendix of the new international classification of headache disorders (ICHD)-3 beta version of headache classification .

Diagnostic criteria The criteria for VM combine the typical signs and symptoms of migraine with the exclusion criteria of other disorders that also elicit vestibular signs . As in migraine without aura, a diagnosis of VM mainly depends on the patient history, for so far there are no clinically useful biomarkers.

Vestibular migraine diagnostic criteria International Bárány Society for Neuro-Otology and the International Headache Society (2012):- A. At least five episodes fulfilling criteria C and D B. A current or past history of migraine without aura or migraine with aura C. Vestibular symptoms of moderate or severe intensity, lasting 5 min to 72 hours D. At least 50 % of episodes are associated with at least one of the following three migrainous features

* Headache with at least two of the following four characteristics

  * Unilateral location
  * Pulsating quality
  * Moderate or severe intensity
  * Aggravation by routine physical activity
* Photophobia and phonophobia
* Visual aura The mechanisms underlying vestibular dysfunction that are related to migraine still need further study and clarification. One explanation proposed is a parallel activation of vestibular and cranial nociceptive pathways.

Experimental studies have demonstrated that trigeminal and vestibular ganglion cells share neurochemical properties and express serotonin, capsaicin, and purinergic receptors. Nociceptive and vestibular afferents with neurochemical similarities converge in brainstem structures like the parabrachial nucleus, the raphe nuclei, and the locus coeruleus. All of these structures play an important role in modulating the sensitivity of pain pathways.

The vestibular rehabilitation become one of the main treatment modalities for patients suffering from vestibular dysfunction, patients are referred for vestibular rehabilitation therapy with aim of helping to relieve them of symptoms of dizziness ,gaze instability, disequilibrium and to improve their functional status.

ELIGIBILITY:
Inclusion Criteria:

* Age: from 20 years to 50 years old.
* Sex: male or female.
* Vestibular migraine

Exclusion Criteria:

1. Evidence of neurological or psychiatric illness.
2. Patients with other types of headache.
3. Evidence of active middle ear disease.
4. History of head trauma, surgery or ototoxic drug therapy
5. Exclude other causes of vestibular disorder

Ages: 20 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: age from age 20 to 50 both male and femele
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
The Role Of Vestibular Rehabilitation Therapy In Management Of Vestibular Migraine Patients | through study completion, an average of 1 year
  quantify the effects of vestibular migrine some of them are as following dizzness handicap inventory

REFERENCES:
- [Background] Headache Classification Committee of the International Headache Society (IHS). The International Classification of Headache Disorders, 3rd edition (beta version). Cephalalgia. 2013 Jul;33(9):629-808. doi: 10.1177/0333102413485658. No abstract available. PMID 23771276